CLINICAL TRIAL: NCT05058079
Title: The Effect of Hand Holding on Patient Satisfaction During for Minimally Invasive Spine Surgery Under Monitored Anesthesia Care. A Single Blinded, Single Center Randomized Controlled Trial
Brief Title: Hand Holding During Light Sedation for Minimally Invasive Spine Surgery Improves Outcomes
Acronym: HHLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1678933
Record Dates: First submitted 2021-09-02; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Spine; Minimally Invasive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-held group (Active Comparator): Patients hand will be held by the anesthesia provider during the procedure. A folded blanket will be over the patient's hand during the procedure and the anesthesia provider will have their hand under the folded blanket holding the patient's hand.
  Interventions: Behavioral: Intraoperative Hand Held
- No hand holding group (No Intervention): No physical contact for comfort or reassurance during the procedure. A folded blanket will be over the patient's hand during the procedure and the anesthesia provider will be next to the patient's hand.

INTERVENTIONS:
Behavioral: Intraoperative Hand Held — Intraoperative hand holding
  Arms: Hand-held group

SUMMARY:
The investigators want to determine whether handholding improves patient satisfaction and reduce patient's anxiety during minimally invasive outpatient spine surgery with monitored anesthesia care.

DETAILED DESCRIPTION:
Minimally invasive spine interventions have emerged as a treatment options for patients with previous spine surgery and patients who have never before been operated upon. These procedures can be done safely in patients with advanced comorbid conditions, previous failed major spine procedures, and in patients who have decided to try the least invasive approach to address their lumbo-sacral spine condition in hopes of avoiding more major and potentially morbid procedures. These endoscopic procedures are typically done as outpatients with light sedation, ideally rendering the patient calm but completely cooperative and able to respond in real-time to questions from the surgeon during the procedure. This has implications for the progress and success of the procedure, the safety of the procedure and allows for a short ambulatory hospital stay.

Hand holding has been shown to improve outcomes such as compliance, procedural success and patient comfort with patients undergoing light sedation for a variety of procedures. The purpose of this study is to determine whether adding hand holding to light sedation for minimally invasive spine procedures has a positive impact on patient satisfaction and perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status 1 to 3
* Outpatient endoscopic spine procedures under light sedation

Exclusion Criteria:

* American Society of Anesthesiology physical status 4 or greater
* Pre-existing neuropathy
* Infection at the site
* Pregnancy
* Patient's refusal or inability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Iowa Satisfaction with Anesthesia Scale (ISAS) | 24 hours after the procedure
  11-item questionnaire designed to measure the satisfaction with monitored anesthesia care. The Iowa Satisfaction with Anesthesia Scale (ISAS) score is the mean of responses to all 11questions. The score can range from a min of -3 to a maximum of +3. The responses are : -3 = disagree very much, -2 = disagree moderately, -1 = disagree slightly, 1 = agree slightly, 2 = agree moderately, and 3 = agree very much. A score of +3 would imply a totally satisfied patient.

SECONDARY OUTCOMES:
Pain Score | Through study completion up to 24 hours after procedure.
  Numerical pain score (0=no pain, 10=worst pain imaginable)
State Trait Anxiety Inventory (STAI) | Before and 24 hours after the procedure
  The 6-item version of the Spielberger 20-item State-Trait Anxiety Inventory (STAI) is a validated short form and correlates well with the standard inventory. It measures state anxiety (how one feels at the moment: "feel questions") and trait anxiety (how one generally feels: "am questions"). It contains six questions with a Likert scale from 1 to 4 (1=not at all, 2=somewhat, 3=moderately so, 4=very much so) The score range is from a minimum of 6 to a maximum of 24. A low score represents no to low anxiety where as a high score represents high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Caiati, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon WA, Lee JW, Seo HK, Oh TH, Park SC, Jeong HJ, Seo IY. Hand-Holding during Cystoscopy Decreases Patient Anxiety, Pain, and Dissatisfaction: A Pilot Randomized Controlled Trial. Urol Int. 2018;100(2):222-227. doi: 10.1159/000485745. Epub 2017 Dec 22. PMID 29275402
- [Background] Dexter F, Candiotti KA. Multicenter assessment of the Iowa Satisfaction with Anesthesia Scale, an instrument that measures patient satisfaction with monitored anesthesia care. Anesth Analg. 2011 Aug;113(2):364-8. doi: 10.1213/ANE.0b013e318217f804. Epub 2011 Apr 25. PMID 21519043
- [Background] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283